CLINICAL TRIAL: NCT04760444
Title: Michigan Men's Diabetes Project (MenD) - Peer Leader Intervention
Brief Title: Michigan Men's Diabetes Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jaclynn Hawkins, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MenD HUM00190932; 2P30AG024824-16 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-18 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Leader Diabetes Self-Management Support (PLDSMS) (Experimental): Participants in the PLDSMS arm will receive 10 hours of group diabetes self-management education (DSME) with a certified diabetes care and education specialist. After the DSME group sessions, the group will complete 6 1-hour weekly diabetes self-management support (DSMS) session led by two peer leaders.
  Interventions: Behavioral: Peer Leader Diabetes Self-Management Support; Behavioral: Virtual Diabetes Self-Management Education
- Control Group (Active Comparator): Participants in the control group will receive 10 hours of group diabetes self-management education (DSME) with a certified diabetes care and education specialist.
  Interventions: Behavioral: Virtual Diabetes Self-Management Education

INTERVENTIONS:
Behavioral: Peer Leader Diabetes Self-Management Support — While the effectiveness of peer-led interventions delivering diabetes-related education and support for short-term clinical, psychosocial, and behavioral improvements is well-established, older Black men in particular are less likely to participate and are at a higher risk of drop-out from these studies. This intervention aims to determine if using older Black men as peer leaders to other older Black men will improve retention rates for this population.
  Arms: Peer Leader Diabetes Self-Management Support (PLDSMS)
Behavioral: Virtual Diabetes Self-Management Education — Participants will attend 10 hours of virtual group diabetes self-management education classes led by a certified diabetes care and education specialist through the online HIPPA compliant Zoom, Med platform.

SUMMARY:
The investigators propose to develop a training for male peer leaders facilitating diabetes self-management education and support (DSMES) to specifically encourage conversations regarding beliefs that affect men's health and to allow modeling of alternative views and perspectives that allow for successful disease management to be framed as competence and strength. Given that the life expectancy for Black men in the US is 71, the investigators hypothesize that targeting men in earlier stages of type 2 diabetes (T2D) will assist greatly in facilitating healthy aging and improving diabetes-related health outcomes later in life.

Based on the investigators previous work, the long-term goal of our research is to determine the most effective, practical, and sustainable approach to provide DSMES to older Black men. The objective is to examine the relative effectiveness, feasibility, and acceptability of a peer-leader DSMES intervention for Black men with T2D. To accomplish this, the investigators will engage in a developmental phase and a validation phase [pilot randomized control trial (RCT)]. The RCT will be conducted with 60 Black adult male residents of metro Detroit, Michigan. Participants will be randomized to a control group or the tailored peer-leader diabetes self-management support group (PLDSMS). All participants will receive DSME with a certified diabetes care and education specialists. Only participants randomized to the PLDSMS group will also receive an additional 6 weeks of DSMS led by the peer leaders. The investigators hypothesize that 1) participants in the PLDSMS group will have improved outcomes (A1c, blood pressure, weight, diabetes distress, self-management behaviors, etc.) over the control group, and 2) an evaluation of measures will confirm efficacy of the PLDSMS.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 55 or older
* Black/African American
* Diagnosis of type 2 diabetes for a six-month duration or longer.

Exclusion Criteria:

* Non-ambulatory
* Serious health conditions (morbid obesity and severe symptomatic heart disease, visual impairment, renal failure, and peripheral neuropathy)
* Psychiatric illness (severity requiring hospitalization)
* Cognitive deficit
* Serious diabetes complications (e.g. blindness) that would impede meaningful participation.

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 25 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclynn Hawkins, MSW, PhD, Principal Investigator — University of Michigan, School of Social Work
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hawkins J, Kloss K, Funnell M, Nwankwo R, Schwenzer C, Smith F, Piatt G. Michigan Men's diabetes project (MenD): protocol for a peer leader diabetes self-management education and support intervention. BMC Public Health. 2021 Mar 22;21(1):562. doi: 10.1186/s12889-021-10613-2. PMID 33752609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Started | 12 | 13
Completed | 11 | 8
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Population: Not all participants came to every health assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 15
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (5.8) | 64.4 (5.6) | 62.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 13 | 25
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25
Hemoglobin A1C [Mean (Standard Deviation); unit: percent Hemoglobin A1C] | 7.7 (2.2) | 7.4 (1.3) | 7.5 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: This outcome measure is change in hemoglobin A1C measured using the DCA 2000 point-of-care testing instrument (value at 3 months minus value at baseline).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: percent of hemoglobin A1c
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
percent of hemoglobin A1c | -0.20 (0.30) | -0.13 (0.31)

2. Primary Outcome: Self-Care Activities
Description: This outcome measure is change in self-care activities as measured by the Summary of Diabetes Self-Care Activities (SDSCA) scale (value at 3 months minus value at baseline). The SDSCA measure is a brief self-report questionnaire of diabetes self-management that includes items assessing the following aspects of the diabetes regimen: general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking. The range for the general diet, specific diet, exercise, blood-glucose testing, and foot care sub scales included below is 0 to 7. Higher scores are indicative of more frequent self-care activities compared to lower scores.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
units on a scale
  General Diet | 1.32 (0.51) | 1.77 (0.98)
  Specific Diet | 0.27 (0.61) | 0.74 (0.49)
  Exercise | 0.95 (0.56) | 2.02 (1.44)
  Blood-Glucose Testing | 0.50 (0.22) | 2.44 (1.89)
  Foot Care | 0.41 (0.53) | 0.04 (0.96)

3. Secondary Outcome: Body Mass Index (BMI)
Description: This outcome measure is change in BMI (value at 3 months minus value at baseline). BMI was calculated using height and weight. Height was measured using a stadiometer. Weight was measured on a high quality, calibrated digital scale. The BMI categories are: Underweight = <18.5; Normal weight = 18.5-24.9; Overweight = 25-29.9; Obesity = BMI of 30 or greater.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
kg/m^2 | -0.31 (0.29) | -0.41 (0.50)

4. Secondary Outcome: Blood Pressure
Description: The outcome measure is the change in blood pressure (value at 3 months minus value at baseline). Blood pressure was measured using the auscultatory method.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
mmHg
  Systolic | -5.23 (2.58) | 10.34 (8.17)
  Diastolic | -1.33 (2.52) | 0.15 (7.3)

5. Secondary Outcome: Depressive Symptom Severity
Description: This outcome measure is change in depressive symptom severity as measured by the Patient Health Questionnaire-2 (PHQ-2) Scale (value at 3 months minus value at baseline). Scores range from 0 to 6. Higher scores are indicative of more depressive symptoms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
units on a scale | -0.45 (0.55) | 0.09 (0.52)

6. Secondary Outcome: Diabetes Self-Efficacy
Description: This outcome measure is change in diabetes self-efficacy as measured by the 8-item Diabetes Self-Efficacy Scale (DSES) (value at 3 months minus value at baseline). The scores for this scale range from 1 to 10. Higher scores are indicative of higher self-efficacy.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
units on a scale | 0.27 (0.48) | 0.33 (0.78)

7. Secondary Outcome: Diabetes Distress
Description: This outcome measure is change in diabetes distress as measured by the 17-item Diabetes Distress Scale (DDS17) (value at 3 months minus value at baseline). Scores for the DDS17 range from 1 to 6. Higher scores are indicate higher diabetes distress. A score of 2 - 2.9 is considered 'moderate distress,' and a score greater than 3.0 is considered 'high distress.'
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
Number analyzed (Participants) | 12 | 13
units on a scale | -3.91 (2.55) | -0.68 (3.28)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Peer Leader Diabetes Self-Management Support (PLDSMS) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
Not all participants were able to go to every health assessment and every support session with the Certified Diabetes Care and Education Specialist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04760444/Prot_SAP_000.pdf